CLINICAL TRIAL: NCT06532643
Title: An Exploratory Clinical Study of Autologous Anti-CD20/CD30 Chimeric Antigen Receptor T Cells (anti-CD20/CD30 CAR-T Cells) in Subjects with Relapsed/Refractory Lymphoma
Brief Title: Safety and Efficacy of Anti-CD20/CD30 CAR-T Cells in Subjects with Relapsed/Refractory Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai First Song Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD20/CD30-CN-A1
Record Dates: First submitted 2024-07-30; First posted 2024-08-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Relapsed/Refractory Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anti-CD20/CD30-CAR-T Cell Therapy (Experimental): Investigational product: anti-CD20/CD30-CAR-T cells Route of administration: Intravenous injection Lymphodepleting chemotherapy regimen: A combination of fludarabine and cyclophosphamide will be administered prior to the infusion of anti-CD20/CD30-CAR-T cells.
  Interventions: Genetic: anti-CD20/CD30-CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: anti-CD20/CD30-CAR-T cells — Each subject will be infused with single dose of anti-CD20/CD30-CAR-T cells. A classic "3+3" dose escalation will be employed.
Drug: Fludarabine — Fludarabine will be given at a dose of 25 mg/m2/day intravenously (IV) for 3 days prior to the infusion of anti-CD20/CD30-CAR-T cells.
Drug: Cyclophosphamide — Cyclophosphamide will be given at a dose of 250 mg/m2/day intravenously (IV) for 3 days prior to the infusion of anti-CD20/CD30-CAR-T cells.

SUMMARY:
This study is an exploratory clinical trial of a single-center, open-label, single-dose treatment of anti-CD20/CD30-CAR-T cells in subjects with relapsed/refractory lymphoma.

DETAILED DESCRIPTION:
The study will enroll subjects with CD20 and CD30-positive lymphoma, CD20-positive lymphoma, or CD30-positive Hodgkin lymphoma. Subjects will receive a single infusion of anti-CD20/CD30-CAR-T cells after screening, PBMC collection, and lymphodepleting chemotherapy. Toxicity will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0) from the National Cancer Institute. Safety of anti-CD20/CD30-CAR-T cell therapy will be evaluated through laboratory tests, including 12-lead electrocardiograms, vital sign checks, etc. Additionally, blood samples will be collected from subjects to study cellular pharmacokinetics and explore the effects of cell therapy on ferritin, C-reactive protein, and related cytokines.

ELIGIBILITY:
Inclusion Criteria

* Patients must meet all of the following criteria to be eligible for the study:

  1. Voluntarily participate in the clinical study. The individual or the legal guardian fully understands the study, sign the informed consent form (ICF), and is willing and able to follow and complete all trial procedures.
  2. Age ≥ 14 years and < 70 years.
  3. Subjects with refractory or relapsed disease after current standard treatments (including allogeneic or autologous hematopoietic stem cell transplantation) who are not suitable for other treatment options, such as a second stem cell transplant. The definitions of relapsed/refractory lymphoma include one of the following situations:

     1. No response to first-line treatment (primary refractory disease, excluding participants intolerant to first-line treatments).

        * Disease progression (PD) as assessed after first-line treatment.
        * Best efficacy of first-line treatment (e.g., 4 cycles of RCHOP) as stable disease (SD), with the duration of SD not exceeding 6 months after the last dose.
     2. No response to second-line or more treatments.

        * PD being the best response to the most recent treatment.
        * Best efficacy of the last line of treatment as SD after at least 2 cycles, with the duration of SD not exceeding 6 months after the last dose.
     3. Refractory after autologous stem cell transplant (ASCT).

        * Disease progression or relapse ≤ 12 months post-ASCT (relapsed patients must have biopsy-proven relapse).
        * If salvage treatment is administered after ASCT, the subjects must not have had a response or relapse after the last line of treatment.
        * Relapsed or refractory disease after two or more lines of systemic treatment.
  4. Lymphoma patients must have target antigens meeting the following criteria:

     1. CD20/CD30 double-positive expressing lymphoma.
     2. Relapse after receiving anti-CD19-CAR-T cell therapy, with CD20 positive lymphoma.
     3. CD20 positive lymphoma that has not previously received anti-CD19-CAR-T cell therapy.
     4. CD30 positive Hodgkin lymphoma.
  5. Subtypes of lymphoma included for enrollment are as follows:

     1. DLBCL-NOS (diffuse large B-cell Lymphoma, not otherwise specified)
     2. Primary mediastinal B-cell lymphoma (PMBCL)
     3. Transformed follicular lymphoma (TFL), previously treated for follicular lymphoma and then transformed to refractory DLBCL
     4. Mantle cell lymphoma
     5. High-grade B-cell lymphoma
     6. Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL)
     7. Hodgkin lymphoma (HL)
  6. ECOG performance status ≤ 2.
  7. Expected survival of at least 12 weeks.
  8. Adequate venous access (for apheresis) and no other contraindications for blood cell separation.
  9. Laboratory tests during screening must meet the following requirements, and the hematological assessment must not have received cell growth factors within 7 days (long-acting colony-stimulating factors (G-CSF/PEG-CSF) require a 2-week interval) or platelet transfusions:

     1. Absolute neutrophil count ≥ 1.0×10^9/L.
     2. Hemoglobin ≥ 60 g/L (without red blood cell transfusion in the last 7 days).
     3. Platelets ≥ 50×10^9/L (unrestricted for CLL indications).
     4. Total bilirubin ≤ 1.5× the upper limit of normal (ULN); or total bilirubin ≤ 3× ULN when the tumor invades liver tissue.
     5. Aspartate transaminase (AST), alanine transaminase (ALT) ≤ 2.5×ULN, with AST/ALT ≤ 5×ULN when the tumor invades liver tissue.
     6. Creatinine < 1.5× ULN and estimated creatinine clearance ≥ 60 mL/min.
  10. Ejection fraction ≥ 45%, with echocardiogram (ECHO) confirming no pericardial effusion (excluding small or physiological amounts), and electrocardiogram results with no clinical significance.
  11. Baseline oxygen saturation > 92% without supplemental oxygen.
  12. Women of childbearing potential must have a negative serum or urine pregnancy test result (women who have undergone surgical sterilization or have been postmenopausal for at least 2 years are not considered of childbearing potential).

Exclusion Criteria:

* Subjects are not eligible to participate in this study if they meet any of the following criteria:

  1. MRI of the brain shows evidence of central nervous system lymphoma; active primary central nervous system DLBL, unless central nervous system involvement has been effectively treated (i.e., participant is asymptomatic), and there has been more than a 4-week gap since local treatment.
  2. Active central nervous system diseases, such as epilepsy, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases with central nervous system involvement.
  3. History of or concurrent diagnosis of malignancies other than CD19+ malignancies.
  4. Clinically significant heart disease or arrhythmias that cannot be controlled with medication.
  5. Presence or suspicion of fungal, bacterial, viral, or other infections that are uncontrolled or require intravenous antibiotics for treatment; uncomplicated urinary tract infections and uncomplicated bacterial pharyngitis are allowed.
  6. Positive for hepatitis B (HBsAg positive and HBV DNA >1000 copies/mL) and hepatitis C (positive for HCV antibodies); syphilis or human immunodeficiency virus (HIV) infection.
  7. Presence of any indwelling catheter or drainage tube (such as percutaneous nephrostomy, indwelling Foley catheter, bile drainage tube, or pleural/peritoneal/pericardial catheter); use of specialized central venous access devices like Port-A-Cath® or Hickman® catheters is allowed.
  8. History of using any of the following medications:

     1. Lenalidomide within 1 day before the apheresis.
     2. Idelalisib (oral PI3Kδ inhibitor) within 2 days before the apheresis.
     3. Short-acting targeted therapy (like tyrosine kinase inhibitors) within 72 hours before the apheresis.
     4. Venetoclax (BCL-2 inhibitor) within 4 days before the apheresis.
     5. Long-acting growth factors (like pegylated filgrastim) within 14 days before the apheresis, or short-acting growth factors or mobilization agents (like G-CSF/filgrastim, plerixafor) within 5 days before the apheresis.
     6. Pharmacological doses of corticosteroids (>5mg/day of prednisone or equivalent doses of other corticosteroids) or other immunosuppressive agents within 7 days before enrollment.
     7. Radiation therapy within 14 days before enrollment.
     8. Systemic cytotoxic drugs, including low-dose maintenance chemotherapy (cyclophosphamide, ifosfamide, bendamustine, methotrexate, or mercaptopurine, vincristine, etc.), within 14 days before enrollment. If bridging therapy is given after apheresis, there should be more than a 7-day gap between bridging therapy and CAR-T cell infusion.
     9. Anti-PD1 or anti-PDL1 within 4 weeks prior to enrollment.
     10. Live vaccines within 4 weeks prior to enrollment.
     11. Donor lymphocyte infusion (DLI) within 4 weeks prior to enrollment.
     12. Immune stimulation or immunosuppressive therapy (like interferon-α, interferon-β, IL-2, etanercept, infliximab, tacrolimus, cyclosporine, or mycophenolate mofetil) within 4 weeks prior to enrollment.
     13. Use of clofarabine or cladribine within 3 months prior to enrollment, or use of PEG-asparaginase within 3 weeks prior to enrollment.
  9. Active graft-versus-host disease (GVHD) rated ≥2 on the CIBMTR acute GVHD grading system or requires systemic steroids at doses greater than physiological levels.
  10. A history of autoimmune diseases in the past 2 years (like Crohn's disease, rheumatoid arthritis, or systemic lupus erythematosus) that has caused damage to end organs or requires systemic immunosuppression/systemic disease-modifying agents.
  11. A history of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant heart diseases within the 12 months prior to enrollment.
  12. A history of genetic syndromes associated with bone marrow failure, such as Fanconi anemia, Kostmann syndrome, or Schwachman-Diamond syndrome.
  13. A history of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation in the 6 months before enrollment. Subjects need to be on preventive anticoagulant medication.
  14. A history of other malignancies (except for non-melanoma skin cancer, in situ breast/cervical cancer, and other malignant tumors that have been effectively controlled without treatment in the past five years).
  15. Use of other investigational medicinal products within 30 days prior to screening.
  16. Pregnant or breastfeeding women of childbearing age. Women who have undergone surgical sterilization or are postmenopausal for at least 2 years are not considered of childbearing potential.
  17. Male and female subjects unwilling to practice contraception from the time they agree to treatment until 12 months after completing the lymphodepleting chemotherapy or CAR-T infusion (whichever is longer).
  18. Any medical activities that could interfere with the safety or efficacy evaluation of the study treatment.
  19. In the judgment of the investigator, subjects are unlikely to complete all required study visits or procedures (including follow-ups) or to comply with the study participation requirements.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerance | 28 days after infusion of anti-CD20/CD30-CAR-T cells
  Incidence of dose-limiting toxicity (DLT)
Manufacturing feasibility | 1 year
  Percentage of subjects for whom the required dose of anti-CD20/CD30-CAR-T cells can be successfully manufactured.

CONTACTS AND LOCATIONS:
Overall Officials: Huaying Ruan, Study Chair — Shanghai First Song Biotechnology Co., LTD; Jian Ge, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No